CLINICAL TRIAL: NCT01228682
Title: A Multi-Centre, Multi-National, Observational Post-Authorisation Safety Study to Document the Drug Utilisation of Samsca and to Collect Information on the Safety of Samsca When Used in Routine Medical Practice
Brief Title: Post-Authorisation Safety Study of Samsca (Tolvaptan) Used in Routine Medical Practice
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-09-101
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: SIADH; Non-SIADH Hyponatremia; Non-Hyponatremia
Keywords: Sodium; SIADH; Hyponatremia; Vasopressin; Salt; Water
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia; Diabetes Insipidus | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who are treated with Samsca.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Samsca 15mg tablet; Samsca 30mg tablet Administration as per Samsca SmPC and medical judgement of treating physician.
  Other Names: Samsca

SUMMARY:
A Drug Utilisation Survey is performed to monitor and document the drug utilisation patterns of Samsca in routine medical practice.

A Post-Authorisation Safety Study is performed to collect information on the safety of Samsca when used in a real-life setting.

DETAILED DESCRIPTION:
Drug Utilisation Survey The drug utilisation analysis will describe the number of prescriptions, their distribution between different medical specialties, and indication for use as compared to the SmPC, patient age and patient gender distributions on a prescription level. In addition, the indication for use will be further categorised as

* SIADH
* Non-SIADH hyponatraemia
* Non-Hyponatraemia

Post-Authorisation Safety Study

Sodium levels at baseline and rate of sodium correction under therapy will be analysed. Safety findings will be described. The number of all non-serious and serious adverse events and the relative frequencies will be analysed in consideration of the risk categories below:

* Renal safety
* Aquaresis-related adverse effects
* Serum sodium correction rate
* Glucose homeostasis
* Cardiovascular safety and hemodynamics
* Respiratory system
* Drug metabolism and drug interactions
* Drug exposure during pregnancy
* Paediatric safety

Subgroup analyses will be performed for all safety findings by indication subgroups (SIADH and other indications), subgroups according to SIADH-underlying diseases, age groups, hepatically impaired patients and renally impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Samsca

Exclusion Criteria:

* Patients who have not signed the data consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are treated with Samsca
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Drug utilisation of Samsca stratified by prescribing medical specialty, indication for use, patient gender and patient age. | 3 years
Samsca sodium correction rates and adverse events in patients treated with Samsca | 3 years

CONTACTS AND LOCATIONS:
Locations (47):
- Denmark (2):
  - Otsuka Study location 45-001, Copenhagen
  - Otsuka Study location 45-006, Holstebro
- Germany (14):
  - Otsuka Study location 49.007, Aachen
  - Otsuka Study location 49.004, Cologne
  - Otsuka Study location 49.016, Dresden
  - Otsuka Study location 49.011, Düsseldorf
  - Otsuka Study location 49.002, Hamburg
  - Otsuka Study location 49.012, Hanover
  - Otsuka Study location 49.018, Hanover
  - Otsuka Study Location 49-020, Heidelberg
  - Otsuka Study location 49-024, Heidelberg
  - Otsuka Study location 49.009, Lübeck
  - Otsuka Study location 49.017, Mannheim
  - Otsuka Study location 49-019, Regensberg
  - Otsuka Study location 49-021, Rostock
  - Otsuka study location 49-001, Würzburg
- Italy (3):
  - Otsuka Study location 39-001, Cuneo
  - Otsuka Study location 39.007, Florence
  - Otsuka Study location 39.005, Siena
- Otsuka Study location 47-001, Lorenskog, Norway
- Spain (8):
  - Otsuka Study location 34-007, Alicante
  - Otsuka Study location 34-014, Castellon
  - Otsuka Study location 34-015, Castellon
  - Otsuka Study location 34-013, Córdoba
  - Otsuka Study location 34-005, Madrid
  - Otsuka Study location 34.017, Majadahonda
  - Otsuka Study location 34-002, Seville
  - Otsuka Study location 34-012, Seville
- Sweden (4):
  - Otsuka Study Location 46.001, Gothenburg
  - Otsuka Study location 46-004, Karlstad
  - Otsuka Study location 46.002, Linköping
  - Otsuka Study location 46-003, Stockholm
- United Kingdom (15):
  - Otsuka Study location 44.024, Birmingham
  - Otsuka Study location 44.019, Coventry
  - Otsuka Study location 44.003, Durham
  - Otsuka Study location 44-023, Hartlepool
  - Otsuka Study location 44.005, Kingston
  - Otsuka Study location 44.006, Liverpool
  - Otsuka Study location 44.016, Liverpool
  - Otsuka Study location 44-001, Manchester
  - Otsuka Study location 44.007, Manchester
  - Otsuka Study location 44.013, Manchester
  - Otsuka Study location 44.021, Nuneaton
  - Otsuka Study location 44-027, Oldham
  - Otsuka Study location 44.015, Oldham
  - Otsuka Study location 44-025, Preston
  - Otsuka Study location 44.004, Southampton

REFERENCES:
- [Derived] Estilo A, McCormick L, Rahman M. Using Tolvaptan to Treat Hyponatremia: Results from a Post-authorization Pharmacovigilance Study. Adv Ther. 2021 Dec;38(12):5721-5736. doi: 10.1007/s12325-021-01947-9. Epub 2021 Oct 25. PMID 34693505